CLINICAL TRIAL: NCT02739100
Title: Pharmacokinetics and Preliminary Bioequivalence of Triferic (Ferric Pyrophosphate Citrate) Administered Via Hemodialysate and Intravenously to Adult CKD-5HD Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rockwell Medical Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RMFPC-16
Record Dates: First submitted 2016-04-11; First posted 2016-04-14 (Estimated); Results first posted 2019-02-01 (Actual); Last update posted 2019-02-01 (Actual); Status verified 2018-08

CONDITIONS: End Stage Renal Disease
Keywords: pharmacokinetics; bioequivalence
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — ferric pyrophosphate; spleen fibrinolytic proteinase (human)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Triferic via Hemodialysate (Experimental): Triferic will be mixed with the liquid bicarbonate concentrate used in the preparation of the hemodialysate solution. This will result in a final Triferic iron concentration in the dialysate of 2 µM (110 µg/L). The patients will receive Triferic via the hemodialysate over the course of the dialysis treatment.
  Intervention Drug: Triferic
  Interventions: Drug: Triferic
- Triferic via IV infusion (Experimental): Patients will receive a single 6.6-mg dose of Triferic iron administered IV over 4 hrs during hemodialysis via the unused heparin infusion line (pre-dialyzer).
  Intervention: Drug: Triferic
  Interventions: Drug: Triferic
- Triferic IV infusion (Experimental): Patients will receive a single 6.6-mg dose of Triferic iron administered IV over 4 hrs during hemodialysis via an infusion port (post-dialyzer).
  Intervention: Drug: Triferic
  Interventions: Drug: Triferic

INTERVENTIONS:
Drug: Triferic
  Other Names: ferric pyrophosphate citrate; FPC

SUMMARY:
The main purpose is to determine the pharmacokinetics (PK) of Triferic iron administered via hemodialysate and via two different intravenous routes in adult patients with chronic kidney disease on chronic hemodialysis (CKD-5HD). It is an open-label, randomized single dose study.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must be able to provide informed consent and have personally signed and dated the written informed consent document before completing any study-related procedures.
2. The patient must have been undergoing chronic hemodialysis for chronic kidney disease for at least 3 months, and is expected to remain on hemodialysis and be able to complete the study.
3. The patient must have a Screening ferritin level of ≥100μg/L.
4. The patient must have a Screening transferrin saturation (TSAT) of 15-45%, inclusive.
5. The patient must have a Screening total iron binding capacity (TIBC) ≥175 μg/dL.
6. The patient must have a Screening hemoglobin (Hgb) concentration ≥9.5 g/dL.
7. The patient must be undergoing hemodialysis at least 3x/week.
8. The patient must have at least a minimally adequate measured dialysis dose defined as single-pool Kt/V (dialyzer clearance of urea multiplied by dialysis time, divided by patient's total body water) ≥1.2, or KIDt/V (online dialyzer clearance measured using ionic dialysance multiplied by dialysis time, divided by patient's total body water) ≥1.2 measured within the 28 days prior to Baseline.
9. Patient is receiving, or can receive anticoagulation for dialysis by a single dose of unfractionated heparin or low molecular weight heparin pre-dialysis; or by intermittent IV heparin bolus.
10. The patient's vascular access for dialysis that will be used during the study must have stable function in the judgment of the Investigator.
11. The patient must agree to discontinue all iron preparations (oral and IV) for 14 days prior to Baseline.
12. Female patients must not be pregnant or breastfeeding. They must have been amenorrheic for the past year or be surgically sterile or agree to not become pregnant by continuous use of an effective birth control method acceptable to the Investigator for the duration of their participation in the study.

Exclusion Criteria:

1. The patient has had an RBC or whole blood transfusion within 4 weeks prior to Screening.
2. The patient requires a continuous infusion of heparin during standard hemodialysis.
3. The patient has had administration of IV or oral iron supplements (including multivitamins with iron) within 14 days prior to Baseline.
4. The patient has known active bleeding from any site other than AV fistula or graft (e.g., gastrointestinal, hemorrhoidal, nasal, pulmonary, etc.).
5. The patient has a living kidney donor identified or living-donor kidney transplant scheduled to occur during study participation. (Note: Patients awaiting deceased-donor transplant need not be excluded.)
6. The patient's vascular access for hemodialysis is a femoral catheter.
7. The patient is scheduled to have a surgical procedure during the study.
8. The patient has had a hospitalization within the 4 weeks prior to Screening (except for vascular access surgery) that, in the opinion of the Investigator, confers a significant risk of hospitalization during the course of the study.
9. The patient has a history of noncompliance with the dialysis regimen in the opinion of the Investigator
10. The patient has a known ongoing inflammatory disorder (other than CKD), such as systemic lupus erythematosus, rheumatoid arthritis, or other collagen-vascular disease, that currently requires systemic anti-inflammatory or immunomodulatory therapy.
11. The patient has any current febrile illness (e.g., oral temperature ≥100.4°F, 38.0°C). (The patient may subsequently become eligible at least 1 week after resolution of the illness.)
12. The patient has known bacterial, tuberculosis, fungal, viral, or parasitic infection requiring anti-microbial therapy or anticipated to require anti-microbial therapy during the patient's participation in this study.
13. The patient is known to be positive for HIV, hepatitis B, or hepatitis C (viral testing is not required as part of this protocol).
14. The patient has cirrhosis of the liver based on histological criteria or clinical criteria (e.g., presence of ascites, esophageal varices, multiple spider nevi, or history of hepatic encephalopathy).
15. The patient has ALT and/or AST levels consistently greater than twice the upper limit of normal at any time during the two months prior to Baseline.
16. The patient currently has any malignancy other than basal or squamous cell skin cancer.
17. The patient has a history of drug or alcohol abuse within the 6 months prior to Screening.
18. The patient participated in an investigational drug study within 30 days prior to Baseline.
19. The patient has any condition that, in the opinion of the Investigator, would make it unlikely for the patient to complete the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-04; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Orlando Clinical Research Center, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: In this cross-over study, all enrolled participants underwent blood sampling over 12 hours for pharmacokinetic (PK) purposes on Day 1. On Days 3, 8, and 10 participants received the following three treatments in a randomized sequence (one treatment per study day): Triferic 2 micromolar via hemodialysate, Triferic 6.6. mg intravenously pre-dialyzer over 3 hours, and Triferic 6.6 mg intravenously post-dialyzer over 3 hours. Blood sampling was conducted over a 12 hour period on each treatment day for PK purposes.
Period: Overall Study
Arm/Group | All Participants
Started | 13
Triferic 2 Micromolar Via Hemodialysate | 13
Triferic 6.6 mg IV Predialyzer | 13
Triferic 6.6. mg IV Post-dialyzer | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Safety Population: All 13 participants completed every arm of the study. Therefore, the baseline demographic characteristics of the Safety Population as a whole also reflect the characteristics of each arm of the study.
Arm/Group | Safety Population
Number analyzed (Participants) | 13
Age, Continuous [Median (Standard Deviation); unit: years] | 49.2 (8.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 12
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 13
Height [Mean (Standard Deviation); unit: centimeters] | 174.3 (9.22)
Weight [Mean (Standard Deviation); unit: kg] | 98.7 (19.34)
C-reactive protein [Mean (Standard Deviation); unit: milligram/deciliter] | .8 (.81)

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK) of Triferic Iron Administered Via Hemodialysate in Adult CKD-5HD Patients: Cmax.
Description: The PK will be done by assessing the mean Cmax of total serum iron from Triferic administered via hemodialysate, compared to Triferic administered at a fixed IV dose of 6.6 mg iron/kg during a single dialysis session.
Time Frame: 1, 2, 3, 4, 5, 6, 8, 10, and 12 hours
Measure: Mean (Standard Deviation); unit: microgram per deciliter
Groups:
- Triferic Via Hemodialysate: Triferic will be mixed with the liquid bicarbonate concentrate used in the preparation of the hemodialysate solution. This will result in a final Triferic iron concentration in the dialysate of 2 µM (110 µg/L). The patients will receive Triferic via the hemodialysate over the course of the dialysis treatment.
  Triferic
- Triferic Via IV Infusion Pre-dialyzer: Patients will receive a single 6.6-mg dose of Triferic iron administered IV over 4 hrs during hemodialysis via the unused heparin infusion line (pre-dialyzer).
- Triferic IV Infusion Post-dialyzer: Patients will receive a single 6.6-mg dose of Triferic iron administered IV over 4 hrs during hemodialysis via an infusion port (post-dialyzer).
Arm/Group | Triferic Via Hemodialysate | Triferic Via IV Infusion Pre-dialyzer | Triferic IV Infusion Post-dialyzer
Number analyzed (Participants) | 13 | 13 | 13
microgram per deciliter | 124 (49.9) | 131 (30.5) | 124 (42.4)

2. Primary Outcome: Pharmacokinetics (PK) of Triferic Iron Administered IV in Adult CKD-5HD Patients: Area Under the Serum Concentration-time Curve From Time Zero to the Time of the Last Quantified Concentration (AUC(Last)).
Description: The PK will be done by assessing the mean area under the serum concentration-time curve from time zero to the time of the last quantified concentration (AUC(last)) and comparing between Triferic administered via hemodialysate and Triferic administered at a fixed IV dose of 6.6 mg iron/kg (pre-dialyzer and post-dialyzer) during a single dialysis session.
Time Frame: 1, 2, 3, 4, 5, 6, 8, 10, and 12 hours
Population: While all subjects were included in PK analysis, some PK samples were below the lower limit of quantitation (BLQ) of the bioanalytical lab assay. Therefore, the number of subjects analyzed differs from the overall total number of study participants.
Measure: Mean (Standard Deviation); unit: hours*microgram/deciliter
Arm/Group | Triferic Via Hemodialysate | Triferic Via IV Infusion Pre-dialyzer | Triferic IV Infusion Post-dialyzer
Number analyzed (Participants) | 12 | 10 | 13
hours*microgram/deciliter | 621 (355) | 630 (275) | 524 (272)

3. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: Safety will be documented by recording the incidence of treatment-emergent adverse events (TEAEs)
Time Frame: 13 days
Population: Safety Population (all enrolled subjects)
Measure: Count of Participants; unit: Participants
Arm/Group | Triferic Via Hemodialysate | Triferic Via IV Infusion Pre-dialyzer | Triferic IV Infusion Post-dialyzer
Number analyzed (Participants) | 13 | 13 | 13
Participants | 1 | 2 | 0

4. Secondary Outcome: Number of Participants With Treatment-emergent Serious Adverse Events (TEAEs)
Description: Safety will be documented by recording the incidence of treatment-emergent serious adverse events (TESAEs)
Time Frame: 13 days
Population: Safety Population (all enrolled subjects)
Measure: Count of Participants; unit: Participants
Arm/Group | Triferic Via Hemodialysate | Triferic Via IV Infusion Pre-dialyzer | Triferic IV Infusion Post-dialyzer
Number analyzed (Participants) | 13 | 13 | 13
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Triferic Via Hemodialysate | Triferic Via IV Infusion Pre-dialyzer | Triferic IV Infusion Post-dialyzer
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 1/13 | 2/13 | 0/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Triferic Via Hemodialysate (N=13) | Triferic Via IV Infusion Pre-dialyzer (N=13) | Triferic IV Infusion Post-dialyzer (N=13)
pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The bioanalytical (ICP MS) assay used for the primary PK analysis was extremely sensitive to hemolyzed samples. The clinical laboratory assay was a better method of quantification for this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days